CLINICAL TRIAL: NCT02730416
Title: ENGOT-EN1/FANDANGO: A Randomized Phase II Trial of First-line Combination Chemotherapy With Nintedanib / Placebo for Patients With Advanced or Recurrent Endometrial Cancer
Brief Title: Combination Chemotherapy With Nintedanib / Placebo in Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other)
Collaborators: North Eastern German Society of Gynaecological Oncology (Other); Belgian Gynaecological Oncology Group (Other); ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENGOT-EN1/FANDANGO
Record Dates: First submitted 2016-01-14; First posted 2016-04-06 (Estimated); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — nintedanib; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Nintedanib (Experimental): Nintedanib 200mg twice daily days 2-21 every 21 days for 6 courses during simultaneous treatment with carboplatin-paclitaxel; afterwards in maintenance 200mg twice daily days 1-21 every 21 days. Treatment continues until progression or unacceptable toxicity.
  Interventions: Drug: Nintedanib or Placebo; Carboplatin, Paclitaxel
- B: Placebo (Placebo Comparator): Placebo twice daily days 2-21 every 21 days for 6 courses during simultaneous treatment with carboplatib-paclitaxel; afterwards in maintenance 200mg twice daily days 1-21 every 21 days. Treatment continues until progression or unacceptable toxicity.
  Interventions: Drug: Nintedanib or Placebo; Carboplatin, Paclitaxel

INTERVENTIONS:
Drug: Nintedanib or Placebo; Carboplatin, Paclitaxel — Arm A: Nintedanib: 200mg orally twice daily d 2-21 q 21 days x 6 courses; afterwards daily dosing, until PD Arm B: Placebo: orally twice daily d 2-21 q 21 days x 6 courses; afterwards daily dosing, until PD In both arms: 6 courses of standard carboplatin and paclitaxel: Carboplatin AUC 5 iv every 21 days; Paclitaxel 175mg/m2 iv every 21 days. Both drugs are continued for maximum six courses or until unacceptable toxicity

SUMMARY:
This study will evaluate the role of addition of an anti-angiogenic agent (Nintedanib/placebo) to conventional combination chemotherapy as concomitant and maintenance treatment in primary advanced or with first relapse of endometrial cancer.

DETAILED DESCRIPTION:
This multicenter, prospective, double-blind, placebo-controlled, randomised phase 2 study is evaluating combination chemotherapy with nintedanib in patients with primary advanced stage (3C2 & 4), or with first relapse of endometrial cancer.

Patients are stratified according to:

1. Stage of disease (stage 3C2 vs. stage 4 vs. recurrent disease)
2. Prior adjuvant chemotherapy (yes/no)
3. Disease status (Measurable disease vs. non-measurable /RECIST 1.1)

Patients are randomized to one of the two treatment arms 1:1 randomization:

* Arm A: Paclitaxel and Carboplatin (6 courses) and Nintedanib (until PD). (Experimental arm)
* Arm B: Paclitaxel and Carboplatin (6 courses) and Placebo (until PD) (Control Arm)

Primary endpoint is PFS. 148 patients to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmed endometrial cancer. (FIGO 2009)

   1. Stage 3C 2
   2. Stage 4 A & B
   3. Relapsed after adjuvant therapy for stage 1-3 disease
2. Patients may have undergone primary surgery.
3. Patients may have received adjuvant chemotherapy for stage 1 - 3.
4. Patients may have received vaginal brachytherapy
5. Patients may have received external beam radiotherapy. Patients who are to be enrolled for stage 3C2 diseases are allowed to receive external beam radiotherapy prior to trial entry.
6. Patients may have received hormonal treatment
7. Patients must have measurable disease or non-measurable disease on CT scan according to RECIST 1.1 outside irradiated field. For stage 3C2 disease patients without measureable or non-measureable disease are accepted.
8. Patients must give informed consent
9. ECOG performance status of 0 -1
10. Patients must have an adequate organ function
11. Life expectancy of at least 12 weeks
12. Patients must be fit to receive combination chemotherapy
13. Patient's age >18 years
14. Patients with preserved reproductive capacity must have a negative pregnancy test (β-HCG test in urine or serum) prior to commencing study treatment

Exclusion Criteria:

1. Sarcomas, small cell carcinoma with neuroendocrine differentiation or non-epithelial cancers.
2. Concurrent cancer therapy
3. Previous Chemotherapy for stage 4 disease or for relapsed disease.
4. Previous treatment with anti-angiogenic/anti VEGF therapy including nintedanib.
5. Concurrent treatment with an investigational agent or participation in another clinical trial.
6. Treatment within 28 days prior to randomisation with any investigational drug, radiotherapy, immunotherapy, chemotherapy, hormonal therapy or biological therapy. Palliative radiotherapy may be permitted for symptomatic control of pain from bone metastases in extremities, provided that the radiotherapy does not involve target lesions, and the reason for the radiotherapy does not reflect progressive disease.
7. Major injuries or surgery within the past 21 days prior to start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period.
8. Relapse within six months after adjuvant chemotherapy (treatment-free interval < 182 days).
9. Previous malignant disease, except patients with other malignant disease, for which the patient has been disease-free for at least three years. Concurrent other malignant disease except for curatively treated carcinoma in situ of the cervix or basal cell carcinoma of the skin.
10. Active infection or other serious underlying medical condition, which might prevent the patient from receiving treatment or to be followed.
11. Evidence of significant medical illness, abnormal laboratory finding or psychiatric illness/social situation that would, in the Investigator's judgement, make the patient inappropriate for this study.
12. Known contraindications to VEGF directed therapy Target Disease Exceptions
13. Known uncontrolled hypersensitivity to the investigational drugs.
14. History of major thromboembolic event defined as:

    * Uncontrolled pulmonary embolism (PE)
    * Deep venous thrombosis (DVT)
    * Other related conditions, though patients with stable therapeutic anticoagulation for more than three months prior randomization are eligible for this study.
15. History of a cerebral vascular accident, transient ischemic attack or subarachnoid haemorrhage within the past 3 months.
16. History of clinically significant haemorrhage in the past 3 months.
17. Radiotherapy to the target lesion within the past 3 months prior to baseline imaging
18. Persistant grade 3 or 4 toxicity from previous chemotherapy and/or radiotherapy, except alopecia. Patients with ongoing ≥ Grade 2 neuropathy are to be excluded.
19. Active brain metastases (e.g. stable for <4 weeks, no adequate previous treatment with radiotherapy, symptomatic, requiring treatment with anti-convulsants; dexamethasone therapy will be allowed if administered as stable dose for at least one month before randomisation).
20. Leptomeningeal disease
21. Significant cardiovascular diseases ( i.e. uncontrolled hypertension, unstable angina, history of infarction within the past 12 months prior to start of study treatment, congestive heart failure > NYHA II, serious cardiac arrhythmia, pericardial effusion) See Appendix 12.
22. Pregnancy or breastfeeding. Patients with preserved reproductive capacity, unwilling to use a medically acceptable method of contraception for the duration of the trial and for 3 months afterwards.
23. Radiographic evidence of cavitating or necrotic tumours with invasion of adjacent major blood vessels.
24. Active or chronic hepatitis C and/or B infection
25. Known hypersensitivity to the trial drugs, or to their excipients.
26. Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug
27. Unable or unwilling to swallow tablets/capsules

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
PFS: Difference in months of Median Progression-Free Survival in experimental arm versus comparator arm | 36 months
  Superiority of Nintedanib arm vs. placebo arm by median PFS increase of 4 months (from 10 months to 14 months) HR: 1.4; power80%; one-sided alpha: 15%. Inclusion period 18 months. Median PFS matures after 14 months of end inclusion

SECONDARY OUTCOMES:
PFS in the sub-populations as described under stratification factors | 32 months
  To be measured (in months) and reported
PFS after consecutive treatment (PFS2). To be measured (in months) and reported | 48 months
  PFS2 is defined along the same timelines as PFS but accounts for the time from randomization to progression or death by any cause on any subsequent line of anticancer therapy.
Disease Specific Survival (DSS) | 48 months
  To be measured (in months) and reported
TSST (Time to Second Subsequent Therapy) | 48 months
  To be measured (in months) and reported
TFST (Time to First Subsequent Therapy) | 48 months
  To be measured (in months) and reported
Overall Survival (OS) | 48 months
  To be measured (in months) and reported
Response Rate (RR). | 32 months
  To be measured (CRs & PRs in %) and reported
Disease Control Rate (DCR) | 32 months
  Disease Control Rate (DCR = Complete Response, Partial Response or Stable Disease for at least 12 weeks). To be measured (CRs, PRs & SDs in %) and reported
Patient Related Outcomes (PROs) | 48 months
  Patient questionnaire results to be presented as as narrative (1-10 scale)
Number of patients with Grade 3 through Grade 5 Adverse Events that are related to study drug. | 36 months
  NCI CTCAE Version 4.0
Compliance in the two treatment arms | 32 months
  Percentage of missed dosages during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor R Mirza, MD, Study Chair — NSGO
Locations (37):
- Belgium (5):
  - Onze Lieve Vrouwziekenhuis, Aalst
  - Cliniques universitaires Saint-Luc, Brussels
  - Antwerp University Hospital, Edegem
  - Ghent University Hospital, Ghent
  - University Hospitals Leuven, Leuven
- Denmark (4):
  - Odense Universitetshospital, Odense, Fyn
  - Aalborg Universitetshospital, Aalborg, Jylland
  - Vejle Sygehus, Vejle, Jylland
  - Rigshospitalet, Copenhagen, Region Sjælland
- Finland (2):
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere
- France (10):
  - Institute Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Léon Bérard Center, Lyon
  - Institut Paoli Calmettes, Marseille
  - ICM (Cancer Institute of Montpellier), Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hospital Group Diaconesses Croix Saint-Simon, Paris
  - Private Hospital Of Côtes D'armor, Plérin
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
- Germany (11):
  - Charité Campus Virchow Clinic, Berlin
  - Klinik Chemnitz gGmbH, Chemnitz
  - University Hospital Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Essen, Essen
  - Kliniken Essen Mitte, Essen
  - Center of Gynecology and Obstetrics, Frankfurt
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - St. Vincentius-Kliniken gAG Frauenklinik mit Hebammenlehranstalt, Karlsruhe
  - Universitätsfrauenklinik Mainz, Mainz
  - Universitätsfrauenklinik am Klinikum Südstadt Rostock, Rostock
  - Universitätsfrauenklinik Ulm, Ulm
- Oslo University Hospital, Oslo, Norway
- Sweden (4):
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Lund
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From January 2024.